CLINICAL TRIAL: NCT01011231
Title: Phase II Study of Gamma-Knife Radiosurgery Using Magnetic Resonance Spectroscopy for Target Definition in Patients With Recurrent Glioma
Brief Title: Study of Gamma-Knife Radiosurgery Using Magnetic Resonance Imaging (MRI) Spectroscopy for Recurrent Glioma
Acronym: GKS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09103
Record Dates: First submitted 2009-11-04; First posted 2009-11-11 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Glioblastoma
Keywords: Gamma Knife radiosurgery; recurrent glioma; MRI; Spectroscopy; Recurrent grade IV glioma (glioblastoma), with two additional exploratory arms for patients with recurrent grade II and grade III gliomas
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Gamma Knife Radiosurgery — Patient treatments will be planned with the Gamma Plan software. The dose will be prescribed to the isodose surface which encompasses the target volume within a range of 50-60% based on a local maximum of 100%. Radiosurgery dose will be prescribed based on volume within the prescribed isodose surface (not to exceed 18 cc)

SUMMARY:
The purpose of this study is to assess the efficacy, of treating patients with recurrent glioblastoma using Gamma-Knife Radiosurgery (GKS) to target a tumor volume defined by a combination of gadolinium enhancement and magnetic resonance spectroscopy (MRS). This is a single center, Phase II trial. A total of 40 glioblastoma patients will be enrolled into the primary arm of the trial. In addition, a minimum of 10 patients with recurrent anaplastic (grade III) gliomas and a minimum of 10 patients with recurrent low-grade (grade II) gliomas will be enrolled into exploratory arms.

The investigators hypothesize that the use of a combination of gadolinium enhancement and elevated Cho:NAA ratio via MRS to determine the treatment target volume for Gamma Knife may be an effective way to treat focally-recurrent glioblastoma.

DETAILED DESCRIPTION:
Study Design: A single-center, single-arm, one-stage phase II clinical trial for patients with recurrent grade IV glioma (glioblastoma), with two additional exploratory arms for patients with recurrent grade II and grade III gliomas.

Patient Numbers: A total of 40 patients with recurrent glioblastoma will be enrolled. In addition, a minimum of 10 patients with recurrent grade III (anaplastic) glioma and a minimum of 10 patients with recurrent grade II (low-grade) glioma will be enrolled independently into separate exploratory arms.

Summary of Patient Eligibility Criteria Histological confirmation of glioma, grades II - IV; prior first-line treatment with surgery, radiotherapy and chemotherapy for malignant (grades III and IV) gliomas; age > 18 years; life expectancy >8 weeks; Karnofsky Performance Status ≥ 60; adequate organ function; signed patient informed consent; willingness to forego additional therapy until evidence of disease progression.

End Points

Primary: Six-month progression-free survival (PFS-6)

Secondary: Median overall survival (mOS), median progression-free survival (mPFS), location of recurrence, symptomatic necrosis rate, reoperation rate, reoperation findings (estimated percentage of viable tumor vs. radiation effect and necrosis), and safety

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, malignant glioma not otherwise specified, low-grade astrocytoma, low-grade oligodendroglioma, low-grade oligoastrocytoma, or low-grade glioma not otherwise specified.
2. Prior first-line treatment with surgery or biopsy followed by fractionated radiotherapy with concurrent temozolomide-containing chemotherapy is required for malignant (grade III or IV) glioma patients. Additional prior chemotherapy is allowed, without limitation on number of recurrences. In patients with low-grade tumors, neither prior radiotherapy nor prior chemotherapy is required.
3. An interval of > 2 months since completion of fractionated radiotherapy.
4. Age > 18 years
5. Life expectancy of at least 8 weeks.
6. Karnofsky Performance Status score (KPS) of ≥ 60
7. Documented recurrent disease: Recurrent disease is defined either as histological confirmation of tumor, as an increase in tumor size of at least 25% based upon serial MR images, or as development of a new site of disease.

   * Tumor size will be calculated using the sum of the largest cross-sectional perpendicular diameters of contrast-enhancing tumor for high-grade tumors, the sum of the largest cross-sectional perpendicular diameters of FLAIR abnormality for low-grade tumors, or as worsened spectroscopic characteristics for any tumor type (development of ≥ 2 new voxels with CNI ≥ 3, or ≥ 25% increase in the sum of the CNI ratios within a group of previously abnormal voxels [where abnormal is defined as CNI ≥ 3]).
   * Disease must be evaluable, but does not need to be measurable.
   * The target site for GKS does not need to be located in a previously-irradiated area.
8. Eligibility for gamma-knife radiosurgery: The decision to treat with gamma-knife radiosurgery will be made by a consensus of the radiation oncology, neurosurgery and neuro-oncology co-chairs or their alternates at the weekly Brain Tumor or Gamma-Knife Tumor Conferences. The MRS defined target volume must be ≤ 15 cc. and not involving eloquent brain (speech/language cortex, motor/sensory cortex, basal ganglia, brainstem, or corpus callosum 2) on an MRI done within 14 days of the planned GKS procedure.
9. BUN < 25 and Cr < 1.7
10. Negative pregnancy test at the time of GKS in any patient who could be pregnant.
11. Willingness to forego additional therapy until evidence of disease progression.
12. Signed and witnessed informed consent and signed authorization for the release of their protected health information.

Exclusion Criteria:

1. MRS defined tumor volume greater than 15 cc.
2. MRS defined tumor volume involving eloquent brain (speech/language cortex, motor/sensory cortex, basal ganglia, brainstem, or corpus callosum).
3. Concurrent treatment with chemotherapy.
4. Active infectious process requiring IV antibiotics.
5. History of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of three years.
6. Other major medical illness judged by the investigator to preclude prolonged follow-up.
7. Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy, as measured by progression-free survival at six months (PFS-6), of treating patients with recurrent glioblastoma using GKS to target a tumor volume defined by a combination of gadolinium enhancement and MRS. | 6 months

SECONDARY OUTCOMES:
To describe PFS and OS in pts with recurrent GBM following GKS targeting a tumor volume defined by a combination of gad enhancement and MRS | 1 year
To further assess the safety of GKS in patients with recurrent glioblastoma | 1 year
To gather initial data regarding the safety and efficacy of treatment of patients with recurrent low-grade or anaplastic glioma with GKS targeting a tumor volume as defined by a combination of gadolinium enhancement and MRS. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Clarke, MD, MPH, Principal Investigator — UCSF Department of Neurosurgery
Locations (1):
- UCSF Department of Neurosurgery, San Francisco, California, United States